CLINICAL TRIAL: NCT05363514
Title: A Pilot Study of Low Dose Naltrexone Use in Patients With Postural Orthostatic Tachycardia Syndrome
Brief Title: Low Dose Naltrexone Use in Patients With POTS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB22-0565
Record Dates: First submitted 2022-05-02; First posted 2022-05-06 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Postural Orthostatic Tachycardia Syndrome
Keywords: POTS; LDN; Low Dose Naltrexone
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome | interventions — Naltrexone; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study drug and placebo will be masked by the pharmacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low Dose Naltrexone (Experimental): Low Dose Naltrexone 4.5mg OD PO. Capsules are masked and provided in blister packs.
  Interventions: Drug: Low Dose Naltrexone
- Placebo (Placebo Comparator): Microcrystalline cellulose 4.5mg OD PO. Capsules are masked and provided in blister packs.
  Interventions: Drug: Microcrystalline cellulose

INTERVENTIONS:
Drug: Low Dose Naltrexone — Participant takes Low Dose Naltrexone 4.5mg PO OD for 120 days. Participant will complete a a 4 week titration to target dose of 4.5mg. Week 1-2: 1.5mg PO OD. Week 3-4: 3.0mg PO OD. Week 5-16: 4.5mg PO OD. Participant will be provided with masked capsules in blister packs.
  Other Names: LDN
  Arms: Low Dose Naltrexone
Drug: Microcrystalline cellulose — Participant takes microcrystalline cellulose 4.5mg PO OD for 120 days. Participant will complete a a 4 week titration to target dose of 4.5mg. Week 1-2: 1.5mg PO OD. Week 3-4: 3.0mg PO OD. Week 5-16: 4.5mg PO OD. Participant will be provided with masked capsules in blister packs.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Many patients with Postural Orthostatic Tachycardia Syndrome (POTS) experience debilitating fatigue and this significantly impacts their daily lives. Unfortunately, there are no treatments to help POTS patients with their fatigue. One medication, called low dose naltrexone (LDN), has been tested as a treatment for fatigue in other medical conditions. In this other research, LDN helped patients feel less fatigue. Other research studies have shown that LDN can help reduce markers of inflammation called cytokines. Reducing these cytokines could help reduce symptoms as well. There have been no research studies testing LDN in POTS to date. We are planning to do a research study to test LDN as a treatment to see if it helps POTS patients feel less fatigue.

DETAILED DESCRIPTION:
Research Objectives: To evaluate LDN as a treatment for fatigue in patients diagnosed with POTS. The primary hypothesis is that LDN will reduce fatigue in patients with POTS when compared to placebo using a 0-100 Fatigue Visual Analogue Scale. The secondary hypotheses are that LDN will improve quality of life in patients with POTS when compared to placebo using the RAND36 Health Related Quality of Life Survey, and that LDN will reduce inflammatory cytokine concentrations in patients with POTS compared to placebo. Tertiary outcomes will compare autonomic symptoms and orthostatic vital signs between LDN and placebo and also evaluate feasibility of a larger scale clinical trial.

Study Design and Methodology: We will recruit 80 patients with POTS across three sites.Participants will be randomized to the LDN group or the placebo group, for a 16 week study. Before beginning the study drug, POTS patients will complete a baseline assessment including fatigue evaluation, cytokine levels, orthostatic vital signs, orthostatic symptoms, and quality of life. After the baseline assessment, POTS patients will begin the study drug titration (LDN or placebo) as follows: 1.5mg for 2 weeks, 3.0mg for 2 weeks, 4.5 mg for 12 weeks. If participants do not tolerate the target dose (4.5mg), then will reduce to the highest tolerable dose. Participants will complete virtual assessments at 1, 2 and 3 months (surveys). Participants will also be provided with a diary to record symptoms. After 4 months, participants will again attend the research clinic/lab for a final assessment (same procedure as the baseline assessment).

Anticipated Outcomes: These data will allow us to evaluate the efficacy of LDN as a treatment in POTS. The results of this study could be used to inform the feasibility and design of larger clinical trials evaluating LDN use in POTS with funding from a national granting agency.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of POTS as defined by the American Autonomic Society consensus statement
* Ability to attend research lab in Calgary, Vancouver or Hamilton, Canada
* Not pregnant and not planning to become pregnant for the duration of the study
* Maintain current other medications at regular doses for the duration of the study

Exclusion Criteria:

* Overt cause for postural tachycardia (e.g. acute dehydration, hyperthyroidism)
* Positive pregnancy test
* Breastfeeding
* Other factors which in the investigator's opinion would prevent participant from completing the protocol, including poor compliance during previous studies
* Current use of Low Dose Naltrexone
* Use of opioid containing medications or positive urine opioid test
* History of alcohol, opioid or other substance use disorder

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Fatigue Visual Analogue Scale (VAS) | 4 months
  Change in Fatigue VAS from pre-treatment (baseline) to treatment (4 months). The score is measured from 0-100 (0 is no fatigue).

SECONDARY OUTCOMES:
RAND 36 Health Related Quality of Life Score | 4 months
  Change in RAND 36 Health Related Quality of Life Score from pre-treatment baseline to treatment (4 months).
Cytokines | 4 months
  Change in plasma cytokine levels from pre-treatment baseline to treatment (4 months)

CONTACTS AND LOCATIONS:
Overall Officials: Satish R Raj, MD MSCI, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dani M, Fedorowski A. Tackling POTS Needs More Than Just a Sympathetic Approach. Hypertension. 2024 Nov;81(11):2248-2250. doi: 10.1161/HYPERTENSIONAHA.124.23716. Epub 2024 Oct 16. No abstract available. PMID 39413203